CLINICAL TRIAL: NCT06573372
Title: A Clinical Validation Study on the Assessment of Sleep Apnea by Smart Watch and Smartphone
Brief Title: Evaluating the Diagnostic Efficacy of Smartwatch and Smartphone for Sleep Apnea
Status: Recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Collaborators: OPPO (Unknown)
Responsible Party: Principal Investigator, Jing MA, Dr., Peking University First Hospital
Other Study IDs: 2024 Research 347-001
Record Dates: First submitted 2024-08-24; First posted 2024-08-27 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Sleep Apnea, Obstructive; smart watch; smartphone; Apnea-Hypopnea Index
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate the diagnostic value of smartphones and watches for OSA screening. The study will be conducted in individuals suspected of having OSA. Subjects will undergo "gold standard" PSG assessment (overnight polysomnography with staff supervision) in a sleep monitoring room, while wearing a smartwatch and smartphone for monitoring. The results will be compared to evaluate the diagnostic value of smartwatches and smartphones for OSA.

DETAILED DESCRIPTION:
OSA is common frequently-occurring disease, in the general population prevalence of 9% to 38%[2] (in apnea hypoventilation index (AHI) 5 for the standard or higher). A OSA, according to the global burden of global nearly 1 billion patients with OSA, and our country is, the most populous country[3] in the OSA sick: on the basis of AHI 5 or more, China has 176 million OSA crowd; With AHI ≥15 as the standard, China has 66 million people with OSA. Although the high prevalence of OSA, diagnostic rate was very low, a study shows there are now about 90% of undiagnosed[4] OSA. The serious influence the diagnosis and treatment of OSA and downstream disease prevention and control.

There are many reasons for the low diagnosis rate of OSA. About the danger of OSA patients with insufficient understanding and OSA diagnosis treatment process link is the more important reason. The OSA diagnosis depends on the patient to the hospital, after outpatient service initiated or portable polysomnography evaluation, limited by registered, see a doctor, make an appointment, monitoring, and many other processes, as well as the level of understanding of OSA patients, many patients with OSA don't want to come to the hospital. With the popularity of intelligent wearable devices, intelligent wearable device can effectively monitor the human multiple physiological indicators, and has high comfort, the cost is low, the detection process is not restricted by time and place, etc. Besides smartphones by smart sensors, collect the snoring, heart shock signals (BCG) and respiratory, physiological parameters, such as non-contact multi-parameter sleep monitoring technology, made possible by the. These are the home sleep monitoring way to provide more convenient and easy to use, makes the risk of OSA screening more convenient[5-8].

The purpose of this study is to evaluate the diagnostic value of smartphones and watches for OSA screening. The study will be conducted in individuals suspected of having OSA. Subjects will undergo "gold standard" PSG assessment (overnight polysomnography with staff supervision) in a sleep monitoring room, while wearing a smartwatch and smartphone for monitoring. The results will be compared to evaluate the diagnostic value of smartwatches and smartphones for OSA.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years; Suspected OSA, scheduled for polysomnography (PSG) Have signed informed consent form.

Exclusion Criteria:

* Co-morbid or definitively diagnosed other sleep disorders, such as central sleep apnea syndrome, narcolepsy, sleepwalking, and insomnia patients with less than 4 hours of nightly sleep; Severe psychiatric or neurological disorders (such as bipolar disorder, schizophrenia, epilepsy, etc.), currently taking sedatives or antipsychotic drugs, or patients with neurological, epileptic, or other disorders causing involuntary movements; Significant somatic disease affecting sleep that has been definitively diagnosed, such as craniocerebral diseases or injuries, pain from various causes, unstable angina, uncontrolled heart failure, persistent atrial fibrillation, or atrial flutter; or patients with implanted pacemakers; Patients who have undergone CPAP titration or treatment Patients with other severe respiratory diseases causing hypoxemia, such as Obesity hypoventilation, severe chronic obstructive pulmonary disease, severe interstitial lung disease, or thoracic restrictive disease; or patients with respiratory failure from various causes; Pregnant or lactating women; Subjects with skin diseases or injuries around the measurement site or allergic to the materials of the research equipment and control device Subjects with either of the following conditions, resulting in the inability to use watch/bracelet-type wearable devices to collect information on both sides of the upper limbs: bilateral limb disability; abnormal skin on the wrist; severe occlusive vascular disease of the upper limbs; significant edema of the upper limbs; skin covering the wrist, such as tattoos, severe hair that covers the skin Subjects whose compliance is judged to be poor or for other reasons deemed unsuitable for participation in by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Suspected OSA patients, scheduled for polysomnography (PSG)
Sampling Method: Non-Probability Sample
Enrollment: 295 (Estimated)
Dates: Start 2024-08-29 (Actual); Primary Completion 2025-03-26 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
diagnostic specificity, sensitivity | 29/8/2024-31/7/2026
  The diagnostic specificity, sensitivity of OPPO smartphone and smartwatch

SECONDARY OUTCOMES:
apnea-hypopnea index (AHI) | 29/8/2024-31/7/2026
  The accuracy of apnea-hypopnea index (AHI) determined by smart watch and smartphones were compared with polysomnography (PSG) .

CONTACTS AND LOCATIONS:
Locations (1):
- Cheng Zhang, Beijing, Beijing Municipality, China